CLINICAL TRIAL: NCT04795180
Title: Pilot Randomized Evaluation of Butyrate Irrigation Before Ileostomy Closure on the Colonic Mucosa in Rectal Cancer Patients: Short-term Outcomes and Microbiota (BUTYCLO)
Brief Title: Pilot Randomized Evaluation of Butyrate Irrigation Before Ileostomy Closure on the Colonic Mucosa in Rectal Cancer Patients (BUTYCLO)
Acronym: BUTYCLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Núria Gómez, MD, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2011043
Record Dates: First submitted 2021-02-22; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Rectal Cancer
Keywords: Ileostomy closure; Butyrate enemas; Microbiota; Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: 1 treatment arm open label
  1 treatment arm double-blind
  1 treatment arm double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-irrigations (No Intervention): No irrigations trough the efferent limb of loop ileostomy
- Butyrate irrigations (Experimental): Butyrate irrigations trough the efferent limb of loop ileostomy
  Interventions: Drug: Irrigations trough the efferent limb of loop ileostomy
- Saline irrigations (Sham Comparator): Saline irrigations trough the efferent limb of loop ileostomy
  Interventions: Drug: Irrigations trough the efferent limb of loop ileostomy

INTERVENTIONS:
Drug: Irrigations trough the efferent limb of loop ileostomy — Irrigations trough the efferent limb of loop ileostomy during 4 weeks previous to ileostomy closure
  Arms: Butyrate irrigations; Saline irrigations

SUMMARY:
Low Anterior resection with total mesorectal excision and diversion loop ileostomy is a gold standard surgical treatment in rectal cancer.

Ileostomy reversal performed in a second stage carries a high burden of postoperative complications.

Terminal ileum and colon dysfunction during bowel disconnection could negatively influence postoperative morbimortality after loop ileostomy reversal in Rectal Cancer patients.

Colonic microflora performs anaerobic breakdown of dietary fibre that reaches the gut in regular patients without ileostomy. One of the short-chain fatty acids (SCFAs) produced by bacteria is butyrate, the preferred substrate to be oxidized by colonocytes.

The effects of butyrate irrigations before ileostomy closure on colonic mucosa will be studied in 45 rectal cancer patients.

The effects of butyrate irrigation trough the efferent limb of loop ileostomy before its closure will be compared to the saline and non-irrigations group.

Short term outcomes, colonic microbiota composition and functional outcomes will be evaluated after ileostomy reversal.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients waiting for an elective ileostomy reversal after Rectal cancer surgical treatment

Exclusion Criteria:

* Inflammatory bowel disease
* Abnormal preoperative findings trough rectoscopy or CT-enema scan that precluded a safe ileostomy closure
* Ileal pouch, poor treatment compliance
* Pregnancy or lactation
* Unwillingness to use adequate contraception throughout the study period
* Combined surgeries
* The impossibility to understand the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-06-21 (Actual)

PRIMARY OUTCOMES:
Postoperative complication rate | Within 90 days after surgery
  Rate of medical and surgical complications within 30 days after surgery using the Dindo-Clavien classification, described as:
  Grade I = Any deviation from the normal postoperative course. Grade 2 = Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Grade III = Requiring surgical, endoscopic or radiological intervention, not under (Grade IIIa) or under general anesthesia (Grade IIIb) Grade IV = Life-threatening complication with single organ (Grade IVa) or Multiorgan dysfunction (Grade IVb) Grade V = Death of a patient.
Length of hospital stay (number of days) | Up to 4 weeks
  Total length of hospital stay will be recorded in days beginning at admission for surgery until discharge.

SECONDARY OUTCOMES:
Diversion colitis evaluation trough rectoscopy in colonic mucosa | At 5-weeks before surgery, At day before surgery
  Diversion colitis was graded as follows: Grade 0: Normal mucosa, Grade 1: Erythematous mucosa, Grade 2: Erythema and mucosa edema and Grade 3: Spontaneous bleeding or bleeding with the slightest contact with rectoscopy
Identification of microbiota modifications in colonic mucosa after irrigations | At 5-weeks before surgery, At day before surgery
  Sequences of the variable portions of the 16s ribosomal RNA gene
Quality of life assessed with Short-Form 36 (SF-36) questionnaire | At hospital discharge and at 1 and 3 months after surgery
  This questionnaire taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/tiredness, and general health perceptions. It also includes a single item that provides an indication of a perceived change in health. Score from 0-100
Anorectal functional outcome assessed by Colorectal Functional Outcome Questionnaire (COREFO) questionnaire | At hospital discharge and at 1 and 3 months after surgery
  Alterations in Colorectal Functional Outcome Questionnaire (COREFO) scores. Score from 0-27

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: Undecided